CLINICAL TRIAL: NCT02734628
Title: A Randomized, Double-blind, Single Center, Intra-individual Comparison Study With Repeated Application to Assess the Wound-healing Efficacy of a 5% Dexpanthenol Ointment Compared With Placebo in Patients With Superficial, Abrasive Wounds
Brief Title: Pilot Study to Assess Number of Patients for Main Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12631; 2006-005508-14 (EudraCT Number)
Record Dates: First submitted 2016-04-07; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Wound Healing
MeSH Terms: interventions — dexpanthenol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexpanthenol (Experimental): A squeeze of ointment, approximately 0.5 cm in length corresponding to an amount of about 0.3 g of ointment, which is equal to 15 mg dexpanthenol , twice daily (once in the morning and once in the evening) over a period of 14 days was applied topically under occluded conditions
  Interventions: Drug: Dexpanthenol (Bepanthen® Wund- und Heilsalbe, BAY81-2996)
- Placebo (Placebo Comparator): Subjects received applications of placebo corresponding to verum
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexpanthenol (Bepanthen® Wund- und Heilsalbe, BAY81-2996) — 30 g of 5% of the active ingredient dexpanthenol plus other ingredients as ointment
  Arms: Dexpanthenol
Drug: Placebo — Placebo to Bepanthen® ointment without active ingredient dexpanthenol
  Arms: Placebo

SUMMARY:
The objective of the study was to investigate the efficacy of Bepanthen® wound healing ointment compared to placebo in a superficial abrasive wound model. The primary objective was the re-epithelization at Day 5.

The secondary objectives were re-epithelization at Days 2, 3, 4, 6, 7, 8, 9, 10 and 15, assessment of cosmetic outcome/acceptance at Day 15 (investigator only) and at Day 36 (investigator and subject), and documentation and analysis of safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian subjects of both genders, 18 to 45 years of age, Fitzpatrick skin type I to IV

Exclusion Criteria:

* Active skin disease, moles, tattoos, strong pigmentation at the test area or scars in the test area that would influence the visual scoring
* History of keloids and hypertrophic scars
* History of plaster sensitivity
* Intake of drugs interfering with the immune system within 30 days before day 1 as well as during the study
* Concomitant therapy with substances affecting blood coagulation within up to 14 days prior to the start of the study as well as during the study
* Any condition or treatment which might influence the study
* Change of hormonal contraception within 3 months prior to enrolment and during the study
* Application of any topical treatment at the test areas during the conduct of the study
* Intensive ultraviolet-light exposure within two weeks before the beginning as well as during the study
* Removal of axillary lymph nodes
* Allergy to the ingredients of the test product
* Pregnancy or lactation
* Any illness on account of which the subject should not participate in the study in the opinion of the investigator
* Psychiatric conditions that might limit the participation in the trial and/or that lead to the assumption that the ability to completely understand the consequences of consent is missing
* Any history of drug addiction or alcoholism in the past 3 years
* Infectious diseases (e.g. hepatitis or AIDS)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2007-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Wound healing effect (=re-epithelization) at Day 5 of the test product and the placebo | At Day 5
  Wound healing effect (=re-epithelization) was determined on the following basis:
  No healing 0% Re-epithelization >0 up to 25% Re-epithelization >25 up to 50% Re-epithelization >50 up to 75% Re-epithelization >75 but not complete Complete closure of surface 100%

SECONDARY OUTCOMES:
Subjective assessment of cosmetic outcome | At Days 15 and 36
  It was assessed by using a visual analog scale (VAS) ranging from 0 being poor, 5 being moderate to 10 being excellent
Number of participants with adverse events | Approximately 5 weeks per subject
Wound healing at Days 2, 3, 4, 6, 7, 8, 9, 10 and 15 after wound induction | At Days 2, 3, 4, 6, 7, 8, 9, 10 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hamburg, Hamburg, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/